CLINICAL TRIAL: NCT02774291
Title: Pilot Study of Adoptive Cell Transfer for the Treatment of Metastatic Cancer That Expresses NY-ESO-1 Using Lymphodepleting Conditioning Followed by Infusion of Anti-NY ESO-1 Murine TCR-Gene Engineered Lymphocytes
Brief Title: Anti-NY ESO-1 mTCR Peripheral Blood Lymphocytes
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Due to lack of accrual the study was formally terminated on 01-JUL-2020. Primary Completion and Study Completion Dates have been revised based accordingly based on respective definitions
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-5254; NCI-2015-01781 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-5254 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Results first posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: HLA-A2 Positive Cells Present; Metastatic Malignant Neoplasm; Metastatic Malignant Neoplasm in the Brain
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — aldesleukin; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (mTCR, aldesleukin) (Experimental): Patients receive standard cyclophosphamide IV over 1 hour on days -7 to -6 and fludarabine phosphate via IVPB over 30 minutes on days -5 to -1 followed by anti-ESO (cancer/test antigen) mTCR-transduced autologous peripheral blood lymphocytes IV over 20-30 minutes on day 0 and aldesleukin IV over 15 minutes approximately every 8 hours on days 0-4. Patients also receive filgrastim SC on days 1-4.
  Interventions: Biological: Aldesleukin; Biological: Anti-thyroglobulin mTCR-transduced Autologous Peripheral Blood Lymphocytes; Drug: Cyclophosphamide; Biological: Filgrastim; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Aldesleukin — Given IV
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Biological: Anti-thyroglobulin mTCR-transduced Autologous Peripheral Blood Lymphocytes — Given IV
  Other Names: Anti-thyroglobulin mTCR-transduced Autologous PBL
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Filgrastim — Given SC
  Other Names: Filgrastim XM02; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tbo-filgrastim; Tevagrastim
Drug: Fludarabine Phosphate — Given IVPB
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; Oforta; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies the side effects of anti-ESO (cancer/test antigen) murine T-cell receptor (mTCR)-transduced autologous peripheral blood lymphocytes and combination chemotherapy with cyclophosphamide and fludarabine phosphate in treating patients with cancer that has spread to other places in the body (metastatic) and expresses the gene NY-ESO-1. Donor white blood cells that are treated in the laboratory with anti-cluster of differentiation (CD)3 may help treat metastatic cancer. Drugs used in chemotherapy, such as cyclophosphamide and fludarabine phosphate, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug (combination chemotherapy) may kill more cancer cells. Aldesleukin may stimulate white blood cells, including natural killer cells, to kill metastatic cancer cells. Giving anti-ESO (cancer/test antigen) mTCR-transduced autologous peripheral blood lymphocytes together with combination chemotherapy and aldesleukin may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of the administration of anti-ESO (cancer/test antigen) mTCR (T cell receptor)-engineered peripheral blood lymphocytes (anti-thyroglobulin mTCR-transduced autologous peripheral blood lymphocytes) plus high-dose aldesleukin following a nonmyeloablative lymphoid depleting preparative regimen in human leukocyte antigen (HLA)-A2 positive patients with metastatic cancer expressing the ESO antigen.

SECONDARY OBJECTIVES:

I. Determine the in vivo survival of T-cell receptor (TCR) gene-engineered cells.

II. Determine the objective response rate by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

OUTLINE:

Patients receive standard cyclophosphamide intravenously (IV) over 1 hour on days -7 to -6 and fludarabine phosphate via intravenous piggy back (IVPB) over 30 minutes on days -5 to -1 followed by anti-ESO (cancer/test antigen) mTCR-transduced autologous peripheral blood lymphocytes IV over 20-30 minutes on day 0 and aldesleukin IV over 15 minutes approximately every 8 hours on days 0-4. Patients also receive filgrastim subcutaneously (SC) on days 1-4.

After completion of study treatment, patients are followed up at 6 weeks, annually for 5 years, and then periodically for 10 years thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Measurable metastatic cancer that expresses NY ESO-1 as assessed by one of the following methods: reverse transcriptase-polymerase chain reaction (RT-PCR) on tumor tissue, or by immunohistochemistry of resected tissue, or serum antibody reactive with ESO
* Confirmation of diagnosis of metastatic cancer by the Laboratory of Pathology at the Montefiore Medical Center
* Patients must have previously received systemic standard care (or effective salvage chemotherapy regimens) for metastatic disease, if known to be effective for that disease, and have been either non-responders (progressive disease) or have recurred
* 3 or fewer brain metastases; Note: if lesions are symptomatic or greater than or equal to 1 cm each, these lesions must have been treated and stable for 3 months for the patient to be eligible
* More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo); Note: patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less or as specified in the eligibility criteria
* Eight weeks must have elapsed from the time of any antibody therapy that could affect an anti-cancer immune response, including anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA 4) therapy, at the time the patient receives the preparative regimen to allow antibody levels to decline; Note: patients who have previously received ipilimumab and have documented gastrointestinal (GI) toxicity must have a normal colonoscopy with normal colonic biopsies
* Willing to sign a durable power of attorney
* Able to understand and sign the informed consent document
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Life expectancy of greater than three months
* Patients must be HLA-A*0201 positive
* Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after cells are no longer detected in the blood
* Serology:

  * Seronegative for human immunodeficiency virus (HIV) antibody; (the experimental treatment being evaluated in this protocol depends on an intact immune system; patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities)
  * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody; if hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be hepatitis C virus (HCV) ribonucleic acid (RNA) negative
* Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus
* Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim
* White blood cell (WBC) >= 3000/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin > 8.0 g/dl
* Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) =< to 2.5 times the upper limit of normal
* Serum creatinine =< to 1.6 mg/dl
* Total bilirubin =< to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl

Exclusion Criteria:

* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant
* Any form of primary immunodeficiency (such as severe combined immunodeficiency disease)
* Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease
* Concurrent opportunistic infections (the experimental treatment being evaluated in this protocol depends on an intact immune system; patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities)
* Concurrent systemic steroid therapy
* History of severe immediate hypersensitivity reaction to any of the agents used in this study
* History of coronary revascularization or ischemic symptoms
* History of or active central nervous system (CNS) or peripheral nerve stimulation (PNS) involvement
* Documented left ventricular ejection fraction (LVEF) of less than or equal to 45%; testing is required in patients with:

  * Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
  * Age >= 60 years old
* Pulmonary function testing in patients with:

  * A prolonged history of cigarette smoking (20 pk/yr of smoking within the past two years)
  * Symptoms of respiratory dysfunction

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira Braunschweig, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (mTCR, Aldesleukin)
Started | 3
Completed | 2
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (mTCR, Aldesleukin)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Toxicity Graded According to NCI-CTCAE Version 4.0
Description: Toxicity graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.0.
Time Frame: Up to 15 years
Population: The study was officially closed on 7/1/2020 as documented on the final progress report dated 8/4/2020. Data for this Outcome Measure limited to 3 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (mTCR, Aldesleukin)
Number analyzed (Participants) | 3
Participants | 2

2. Secondary Outcome: Number of Participants Demonstrating in Vivo Survival of TCR Gene-engineered Cells
Description: TCR and vector presence will be quantitated in PBMC samples (5-10mL) using established PCR techniques. This will provide data to estimate the in vivo survival of lymphocytes derived from the infused cells. In addition, measurement of CD4+ and CD8+ T-cells will be conducted and studies of these T-cell subsets in the circulation will be determined by using specific PCR assays capable of detecting the unique DNA sequence for each retroviral vector engineered T-cell. Descriptive statistics will be used to determine the in vivo survival of TCR gene-engineered cells.
Time Frame: 6 weeks post evaluations scan and at 3, 6, and 12 months and annually thereafter
Population: Data was never collected/aggregated and in vivo survival of TCR gene-engineered cells outcome measure was never analyzed due to the limited number of participants and early termination. The study was officially closed on 7/1/2020 as documented on the final IRB progress report dated 8/4/2020.
Arm/Group | Treatment (mTCR, Aldesleukin)
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants Demonstrating Objective Response Rate (Complete Response + Partial Response) Using RECIST Criteria
Description: Objective Response Rate will be graded based on the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 criteria.
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study
  Descriptive statistics will be used to determine the objective response rate.
Time Frame: Up to 15 years
Population: Data to support the Objective Response Rate outcome measure was never collected and analyzed due to the limited number of participants enrolled and early termination. The study was officially closed on 7/1/2020 as documented on the final progress report dated 8/4/2020.
Groups:
- Treatment (mTCR, Aldesleukin): Patients receive standard cyclophosphamide IV over 1 hour on days -7 to -6 and fludarabine phosphate via IVPB over 30 minutes on days -5 to -1 followed by anti-ESO (cancer/test antigen) mTCR-transduced autologous peripheral blood lymphocytes IV over 20-30 minutes on day 0 and aldesleukin IV over 15 minutes approximately every 8 hours on days 0-4. Patients also receive filgrastim SC on days 1-4.
  Aldesleukin: Given IV
  Anti-thyroglobulin mTCR-transduced Autologous Peripheral Blood Lymphocytes: Given IV
  Cyclophosphamide: Given IV
  The study was closed via final progress report on 08/03/2020, no new data are available.
  Filgrastim: Given SC
  Fludarabine Phosphate: Given IVPB
  Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Treatment (mTCR, Aldesleukin)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 9 months
Description: The study was closed via final progress report on 08/03/2020 and no further AE data were collected.
Arm/Group | Treatment (mTCR, Aldesleukin)
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (mTCR, Aldesleukin) (N=3)
Headache (Nervous system disorders) | 2 — Intermittent, Grades 1-2
Edema limbs (General disorders) | 1 (2) — Bilateral legs, right>left. Grade 2
Weight Gain (Investigations) | 2 (2) — Grade 1
Diarrhea (Gastrointestinal disorders) | 1 — Intermittent, highest severity Grade 2
Vomiting (Gastrointestinal disorders) | 2 — Intermittent, Grades 1-2
Nausea (Gastrointestinal disorders) | 1 — Intermittent, highest severity Grade 2
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) — Right Lower Extremity, Grade 1
Chills (General disorders) | 2 (2) — Grade 1
Hypotension (Vascular disorders) | 2 — Intermittent, highest severity Grade 2
Sinus Tachycardia (Cardiac disorders) | 1 — Intermittent, highest severity Grade 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1 — Intermittent, highest severity Grade 2
Neutrophil Count Decreased (Investigations) | 2 — Intermittent, Grades 2-4
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) — Intermittent,, Grades 1-2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — At rest, Grade 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 — Intermittent, highest severity Grade 1
Lethargy (Nervous system disorders) | 1 (1) — Grade 1
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Generalized, abdomen-back. Grade 1
Confusion (Psychiatric disorders) | 1 (1) — Grade 1
Fatigue (General disorders) | 1 (1) — 'generalized weakness', Grade 1
Fever (General disorders) | 1 (1) — Grade 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 — Intermittent, Grades 1-3
Creatinine Increased (Investigations) | 1 (1) — Grade 1
Platelet Count Decreased (Investigations) | 1 (1) — Grade 4
Chest Pain (General disorders) | 1 (1) — Nonspecific. Grade 2
Flushing (Vascular disorders) | 1 (1) — Grade 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Jaw, Grade 2
Appetite (Metabolism and nutrition disorders) | 1 (1) — Loss of appetite. Grade 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 — Intermittent, positional desaturation (lying down). Grade 2
Acidosis (Metabolism and nutrition disorders) | 1 (1) — Grade 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) — Grade 4
Blood Bilirubin Increased (Investigations) | 1 (1) — Grade 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 2
Urinary Frequency (Renal and urinary disorders) | 1 (1) — Grade 1
Tachycardia (Cardiac disorders) | 1 (1) — Nonspecified, Grade 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 — Intermittent, Grade 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) — 'hair loss.' Grade 1
Mucositis oral (Gastrointestinal disorders) | 1 (1) — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT02774291/Prot_SAP_000.pdf